CLINICAL TRIAL: NCT07330856
Title: Evaluation of Treatments for Recent Dry or Productive Cough Accompanying Benign Viral Rhinopharyngeal Infectious Episodes.
Brief Title: Evaluation of Treatments for Dry or Productive Cough
Acronym: SPRATO
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RBHP 2025 PICKERING 2; 2025-A02027-42 (Other: IDRCB)
Record Dates: First submitted 2025-12-19; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Cough
MeSH Terms: conditions — Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group CDN (Experimental): VB-ChSp-D-N® (CDN) is a film-forming liquid dressing designed for the treatment of cough.
  Interventions: Combination Product: Group CDN
- Group CW (Experimental): VB-ChSp-W® (CW) is a film-forming liquid dressing designed for the treatment of cough.
  Interventions: Combination Product: Group CW

INTERVENTIONS:
Combination Product: Group CDN — VB-ChSp-D-N® (CDN) is a film-forming liquid dressing designed for the treatment of cough. Key Features: *Administration: - Initial Dose (Day 1): 4 sprays every 30 minutes for 2 hours, then 4 sprays every 3-4 hours for the remainder of the day. - Maintenance Dose (Days 2-7): 4 sprays every 3-4 hours (4 times daily) *Mechanism: Forms a protective film that draws fluid from the tissues, creating an outward flow. This lifts contaminants from the throat's surface and ensures sustained hydration, thereby alleviating cough. *Use Case: Targeted Throat Cough Relief. Additional Notes: *Non systemic (local action). *CE-marked as a Class I medical device (under EU Directive 93/42/EEC).
  Arms: Group CDN
Combination Product: Group CW — VB-ChSp-W® (CW) is a film-forming liquid dressing designed for the treatment of cough. Key Features: *Administration: - Initial Dose (Day 1): 4 sprays every 30 minutes for 2 hours, then 4 sprays every 3-4 hours for the remainder of the day. - Maintenance Dose (Days 2-7): 4 sprays every 3-4 hours (4 times daily) *Mechanism: Forms a protective film that draws fluid from the tissues, creating an outward flow. This lifts contaminants from the throat's surface and ensures sustained hydration, thereby alleviating cough. *Use Case: Targeted Throat Cough Relief Additional Notes: *Non systemic (local action) *CE-marked as a Class I medical device (under EU Directive 93/42/EEC).
  Arms: Group CW

SUMMARY:
This is a post-marketing, monocentric, open-label, randomized, two-arm, parallel-group clinical study. Its primary objective is to evaluate the real-world tolerability and safety profile of two CE-marked Class I medical devices formulated as throat sprays: VB-ChSp-D-N (CDN) and VB-ChSp-W (CW), when used for symptomatic relief of cough associated with suspected viral upper respiratory infections.

The study is designed as a Category 4.2 clinical investigation according to applicable regulations, focusing on devices already bearing the CE mark and used within their intended purpose as per the manufacturer's instructions. The hypothesis is that both devices demonstrate an acceptable real-world tolerability profile, with a pre-defined threshold for adverse event incidence not to be exceeded, while also showing a positive impact on cough symptoms and patient quality of life.

Methodological Framework:

Design: A two-stage Fleming design will be implemented separately for each device arm to sequentially assess the primary tolerability outcome. This design allows for an early stopping rule if an unacceptable number of adverse events is observed in the first cohort of participants.

Population: The study will enroll adult patients (aged 18-65) presenting with an acute cough of less than three weeks' duration, attributed to a suspected viral etiology (e.g., common cold, viral pharyngitis). Key exclusion criteria are in place to ensure a population suitable for device evaluation, including the absence of underlying chronic respiratory conditions, bacterial infection, or use of prohibited medications that could confound results.

Intervention: Eligible participants will be randomized in a 1:1 ratio to use either the CDN spray (n ≤ 29) or the CW spray (n ≤ 29) according to the prescribed labeling for a 7-day treatment period.

Assessments: Data collection emphasizes real-world evidence capture. Participants will use an electronic daily diary throughout the treatment period to report cough symptoms (via a validated patient-reported outcome instrument), any adverse events, concomitant medications, and potential device defects (recorded as a binary yes/no occurrence). Additionally, patient-reported quality of life related to cough will be assessed using a standardized questionnaire at baseline (Day 1) and at the end of treatment (Day 8). Two on-site clinical visits (Days 1 and 8) will be conducted for clinical examination and procedures.

Outcome Measures:

The study employs a hierarchical assessment of endpoints:

Primary Outcome: Tolerability/Safety, defined by the incidence of device-related adverse events collected via the electronic diary.

Key Secondary Outcome: Clinical Efficacy, measured by the change from baseline in the Total Cough Symptom Score (TCSS).

Other Secondary Outcomes: These include the impact on cough-specific quality of life domains (sleep, daily activities, fatigue, irritability) and the incidence of device malfunctions or use errors.

The study will be conducted at a single investigational site (Clermont-Ferrand University Hospital, France).

ELIGIBILITY:
Inclusion Criteria:

* Male or female,
* Aged 18 to 65 years,
* Presenting with an acute dry or productive cough for less than 3 weeks, associated with one of the following viral conditions: Acute viral rhinitis, Acute viral rhinopharyngitis, Acute viral tonsillitis, Acute viral pharyngitis / tonsillitis,
* For patients with suspected pharyngitis/tonsillitis: McIsaac score < 2 or a negative rapid antigen detection test for Group A beta-hemolytic Streptococcus,
* Effective contraception for female patients of childbearing potential,
* Sufficient cooperation and understanding to comply with the requirements of the trial,
* Acceptance of registration in the SI-RIPH database (Système d'Information pour la Recherche sur les Produits de Santé),
* Having received clear information and agreeing to provide written informed consent,
* Covered by the French national health insurance system

Exclusion Criteria:

* Hypersensitivity or history of allergy to any component of the investigational products,
* Severe, poorly tolerated cough,
* Complicated acute rhinitis (e.g., acute bacterial sinusitis, acute otitis media, acute bronchitis, or pneumonia),
* Chronic or allergic rhinosinusitis,
* Bacterial tonsillitis or pharyngitis,
* Positive antigen test for influenza A/B or COVID-19 requiring etiological treatment per current guidelines (Appendix 5),
* Concurrent use of antitussives, bronchodilators, inhaled corticosteroids, other pulmonary-targeted therapies, or medications known to induce cough (such as ACE inhibitors, ARBs, etc.), antibiotics, antivirals, or any other treatment deemed incompatible with the study by the investigator,
* Recent ENT surgery (<6 months),
* Pulmonary disease (e.g., COPD, asthma),
* Immunodeficiency (based on patient declaration),
* Comorbidities or a health status judged incompatible with the trial by the investigator (e.g., Gastroesophageal Reflux Disease [GERD] or abnormal lung auscultation),
* Pregnant or breastfeeding women,
* Regular tobacco smoker (as judged by the investigator),
* Current participation in another clinical trial, being in an exclusion period from a previous trial, or having received total compensation exceeding 6000 euros in the 12 months prior to study start,
* Under legal protection measures (guardianship, trusteeship, deprivation of liberty, judicial safeguard).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Collection of adverse events (AEs) during the use of investigational products CDN and CW recorded in an electronic daily diary. | From visit 1 (Day 1) and Visit 2 (Day 8)

SECONDARY OUTCOMES:
Total Cough Symptom Score | At Visit 1 and from day 5 to day 7
  Clinical improvement (yes/no), defined as a reduction of at least 30% in the Total Cough Symptom Score from its baseline value to the average of scores measured during the last 3 days of product use (Days 5, 6, and 7).
  Details of Total Cough Symptom Score (TCSS) is composed of 9 items (ranging from 0 to 90):
  * Frequency of cough
  * Severity of cough
  * Coughing fits / Paroxysmal cough
  * Chest or abdominal pain due to coughing
  * Hoarse voice due to coughing
  * Shortness of breath due to coughing
  * Sore throat sensation
  * Interruption of conversations (in person or on the phone) due to coughing
  * Difficulty falling asleep due to coughing
Sleep measurement | From Visit 1 (Day 1) to Visit 2 (Day 8)
  Change in quality of sleep measured before (Day 1) and after (Day 8). Participants will indicate their level of discomfort on a Visual Analog Scale ranging from 0 ("not at all bothersome/impacted") to 10 ("extremely bothersome/severely impacted").
Daily activities measurement | [Time Frame: From Visit 1 (Day 1) to Visit 2 (Day 8)]
  Change in daily activities measured before (Day 1) and after (Day 8). Participants will indicate their level of discomfort on a Visual Analog Scale ranging from 0 ("not at all bothersome/impacted") to 10 ("extremely bothersome/severely impacted").
Fatigue measurement | [Time Frame: From Visit 1 (Day 1) to Visit 2 (Day 8)]
  Change in fatigue measurement measured before (Day 1) and after (Day 8) product use. Participants will indicate their level of discomfort on a Visual Analog Scale ranging from 0 ("not at all bothersome/impacted") to 10 ("extremely bothersome/severely impacted").
Irritability measurement | [Time Frame: From Visit 1 (Day 1) to Visit 2 (Day 8)]
  Change in irritability measurement measured before (Day 1) and after (Day 8) product use. Participants will indicate their level of discomfort on a Visual Analog Scale ranging from 0 ("not at all bothersome/impacted") to 10 ("extremely bothersome/severely impacted").
Collection of defects in products | From Visit 1 (Day 1) to Visit 2 (Day 8)
  Device defects were monitored through a binary (yes/no) reporting system in an electronic daily diary.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Clermont-ferrand, Clermont-Ferrand, France